CLINICAL TRIAL: NCT01538914
Title: A Comparison Between the Analgesic Effect of Intravenous Patient-controlled Analgesia and of Paravertebral Block After Video Assisted Thoracoscopic Surgery
Brief Title: Analgesic Effect of Intravenous Patient-Controlled Analgesia (IV PCA) Versus Paravertebral Block After Video Assisted Thoracic Surgery (VATS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JHBahk_VATS PVB
Record Dates: First submitted 2012-02-16; First posted 2012-02-24 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Postoperative Pain After Video Assisted Thoracic Surgery
MeSH Terms: interventions — Passive Cutaneous Anaphylaxis

ARMS (2):
- PVB (Experimental): Postoperative pain is controlled with local analgesics delivered via PVB.
  Interventions: Procedure: paravertebral block
- PCA (Active Comparator): Postoperatve pain is controlled with intravenous PCA.
  Interventions: Procedure: PCA

INTERVENTIONS:
Procedure: paravertebral block — Postoperative pain is controlled with local analgesics via PVB.
  Arms: PVB
Procedure: PCA — Postoperative pain is controlled with intravenous PCA.
  Arms: PCA

SUMMARY:
The purpose of this study is to compare the analgesic effect of paravertebral block with that of intravenous patient-controlled analgesia after video assisted thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving video assisted thoracic surgery

Exclusion Criteria:

* patients with cardiovascular disease
* patients with neurologic disease
* patients with contraindications to paravertebral block or epidural block
* patients with history of previous VATS
* patients with pain at the expected incision site

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-02; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
severity of acute postoperative pain when moving | 24 hours after VATS

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea